CLINICAL TRIAL: NCT00662584
Title: The Efficacy of Functional Magnetic Resonance Imaging (fMRI) Guided Low Frequency Repetitive Magnetic Transcranial Stimulation (rTMS) Therapy on Symptoms of Generalized Anxiety Disorder (GAD)
Brief Title: Repetitive Magnetic Transcranial Stimulation (rTMS) in the Treatment of Generalized Anxiety Disorder (GAD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Phillis and Brian Harvey Foundation (Unknown); Saban Family Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-05-045-01
Record Dates: First submitted 2008-04-14; First posted 2008-04-21 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Generalized Anxiety Disorder
Keywords: repetitive magnetic transcranial stimulation (rTMS); functional magnetic resonance imaging (fMRI)
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): This was an open-label study - all subjects received the intervention (rTMS treatment)
  Interventions: Procedure: Repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Procedure: Repetitive transcranial magnetic stimulation (rTMS) — transcranial magnetic stimulation (TMS) at .5 HZ for 20s

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) is a noninvasive method that holds promise for treating several psychiatric disorders. Yet the most effective location and parameters for treatment need more exploration. Also, whether rTMS is an effective treatment for individuals with a DSM-IV diagnosis of Generalized Anxiety Disorder (GAD) has not been empirically tested. The goal of this pilot study is to evaluate whether fMRI guided rTMS is effective in reducing symptoms of GAD.

DETAILED DESCRIPTION:
This study utilized a 3-week open-label design to evaluate the efficacy of fMRI guided rTMS in the treatment of GAD.

We first used functional magnetic resonance imaging (fMRI) during the gambling task to localize anxiety-related brain activations in each individual participant, and then used this information to guide treatment with repetitive transcranial magnetic stimulation (rTMS).

TMS was delivered to the target site at a frequency of 1 Hz for 20 minutes (900 total pulses). The intensity of the TMS was set to 90% of the passive motor threshold for each participant.

The primary efficacy measures include the Clinical Global Impression of Improvement (CGI-I) and the Hamilton Anxiety Rating Scale (HARS). Response to treatment was defined as a reduction of 50% or more on the HARS and symptom remission was defined as a CGI-I score of 1 or 2 ("much improved" or "very much improved" respectively) and a score ≤ 8 on the HARS. Data was entered anonymously into an Excel spreadsheet and analyzed by the UCLA Semel Institute Statistical Core. The analysis was done on the intent to treat sample using last observation carried forward (LOCF). A one-sample paired t-test was used to compare endpoint to baseline means on the HARS, with a significance level set at p= 0.05, two-tailed.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female outpatients age 18 to 65 years, inclusive
* The subject meets DSM-IV criteria for Generalized Anxiety Disorder as determined by the MINI.
* Sexually active female patients of childbearing potential must be practicing at least one or more the following methods of contraception during the study: intrauterine device (IUD), barrier method in combination with a spermicide, oral/hormonal contraception or abstinence. Female patients of childbearing potential must have a negative pregnancy test prior to receiving study drug.
* Written informed consent must be obtained from the subject prior to study participation.
* The subject is in good medical health or with chronic medical conditions which are currently stable.
* No current abuse of alcohol or other substance.
* The subject has a total score of 20 or more on the SIGH-A at screening.
* The subject has a Clinical Global Impression (CGI) Severity score of 4 or more at screening.

Exclusion Criteria:

* The subject meets DSM-IV criteria for an Axis I diagnosis (other than GAD) as the primary diagnosis (i.e., schizophrenia, mood disorder, psychosis, anorexia nervosa) as determined by the MINI.
* The subject is clinically judged by the investigator to be at risk for suicide or is acutely suicidal as objectively measured by the MINI and MSE.
* The subject is clinically judged by the investigator to be at risk for homicide or is acutely homicidal as objectively measured by the MINI and MSE.
* The subject has a psychiatric condition that would require inpatient, or partial psychiatric hospitalization.
* Seizure disorders.
* Significant history of medical disease (i.e. cardiovascular, hepatic (e.g. cirrhosis, hepatitis B or C) renal, gynecological, musculoskeletal, neurological, gastrointestinal, metabolic, hematological, endocrine, cancer with a metastatic potential or progressive neurological disorders) which could impair reliable participation in the trial or necessitate the use of medication not allowed by this protocol.
* The subject is pregnant, planning to become pregnant, or nursing. If a subject becomes pregnant, she will be discontinued immediately and followed appropriately.
* Concomitant therapy with another investigational drug, or participation in an investigational drug study within one month prior to entering this study.
* Current psychotherapeutic treatment except for treatment with Specific Reuptake Inhibitor (SSRIs) medications which include: Fluoxetine (Prozac), Paroxetine (Paxil), Sertraline (Zoloft), Luvox (Fluvoxamine), and Citalopram. Potential subjects may remain on one of the SSRI medications provided that he or she has been on a stable dose for at least 4 weeks prior to entering this study; this dose remains stable throughout the remainder of this study; and it can be determined that this medication is not exacerbating the anxiety symptoms.
* History of poor compliance or in the Investigator's judgment patients any subject whose treatment as an outpatient would be clinically contraindicated
* The subject has attempted suicide one or more times within the past twelve months
* The subject has a Structured Hamilton Depression Rating Scale (SIGH-D) score above 38 which suggests a moderate to severe clinical level of depressive symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-08; Primary Completion 2007-03 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Structured Interview for the Hamilton Anxiety Rating Scale (SIGH-A) | Week 0, 3, 6
The Clinical Global Impression (CGI) Scale of Severity/Improvement | Week 0, 3, 6

SECONDARY OUTCOMES:
Structured Interview for the Hamilton Depression Rating Scale (SIGH-D) | Week 0 and 6
The Side-Effects Questionnaire | Week 0, 3, 6

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Bystritsky, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States